CLINICAL TRIAL: NCT02033538
Title: A Phase II Trial of Neoadjuvant Chemotherapy With Nanoparticle Albumin-bound Paclitaxel and Fluorouracil Followed by Surgery in Patients With Locally Advanced Squamous Cell Carcinoma of Esophagus
Brief Title: Neoadjuvant Chemotherapy of Nanoparticle Albumin-bound Paclitaxel in Squamous Cell Carcinoma of Esophagus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This clinical trial was closed due to slow recruitment of patients.
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Qiong Zhao, Chief of Department of Thoracic Oncology, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYTOP1403
Record Dates: First submitted 2013-12-16; First posted 2014-01-10 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Squamous Cell Carcinoma of Esophagus
Keywords: Neoadjuvant chemotherapy; Nab-Paclitaxel; Carcinoma of Esophagus
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — Taxes; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nanoparticle albumin-bound paclitaxel (Experimental): Paclitaxel protein-bound particles for injectable suspension (albumin-bound) 125 mg/m2 (IV over 30 min) (days 1 and 8) on 21 day cycle
  Interventions: Drug: nanoparticle albumin-bound paclitaxel

INTERVENTIONS:
Drug: nanoparticle albumin-bound paclitaxel — Paclitaxel protein-bound particles for injectable suspension (albumin-bound) 125 mg/m2 (IV over 30 min) (days 1 and 8) on 21 day cycle
  Other Names: nab-paclitaxel

SUMMARY:
Albumin-bound paclitaxel regimen in advanced NSCLC has a better tumor response rate and safety than solvent-based paclitaxel. However, the safety and efficacy is uncertain in neoadjuvant therapy in esophageal cancer. The objective of this single-arm phase II trial was to evaluate the benefit of neoadjuvant chemotherapy with nanoparticle albumin-bound paclitaxel plus 5-fluorouracil in patients with locally advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
In the past decade, clinical trials have evaluated the role of neoadjuvant chemotherapy, radiation, or both, for patients with surgically resectable esophageal carcinoma, but have all failed to demonstrate a consistent survival benefit. In Eastern countries, preoperative chemotherapy followed by radical surgery became one of the treatment strategies for resectable, clinical stage II or III esophageal cancer. In an effort to improve the efficacy of systemic chemotherapy, we conducted a prospective study to evaluate the regimen of nanoparticle albumin-bound paclitaxel plus 5-fluorouracil as perioperative therapy for patients with resectable esophageal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the thoracic esophagus, including the gastroesophageal junction (Siewert type I)
* Locally advanced disease that is technically operable with curative intent (R0)
* T3, N0 OR T1-3, N+ OR T4, Nx
* No T1-2, N0
* No inoperable T4 (unequivocal organ involvement)
* No distant metastasis, including M1a lymph node status
* Lymph nodes suspicious of M1a status by CT scan, PET scan, or ultrasound must be verified by fine-needle aspiration cytology
* No carcinoma of the cervical esophagus
* Obstructive tumors allowed

Exclusion Criteria:

* Not suitable to surgery
* cervical Esophageal Carcinoma(distance of incisor tooth<19cm)
* early Esophageal Carcinoma(Stage I)
* complete esophageal obstruction，Esophageal perforation or hematemesis
* other malignant tumors, except for skin basal cell carcinoma, or cervical carcinoma in situ
* pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives
* Uncontrolled seizures or psychiatric diseases, loss of control over their own behavior
* History of serious allergic or castor oil allergy
* Patients who are not suitable to participate in the trial according to researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
response rate | From date of treatment until the date of progression, assessed up to 2 months
  pathological response rate and clinical response rate

SECONDARY OUTCOMES:
Overall survival | Overall survival was measured from the date of treatment to the date of death, or last follow-up,assessed up to 48 months
Progression-free survival | Progression-free survival was measured from the date of treatment to the date of first evidence of relapse or death due to any cause,assessed up to 36 months
Adverse events | During the chemotherapy,an expected average of 3 weeks
  Adverse events were classified according to U.S. National Cancer Institute common toxicity criteria, version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Zhao, MD, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The first affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China